CLINICAL TRIAL: NCT01950507
Title: Evaluation of Serum Concentrations of Budesonide in Patients Treated for Gastrointestinal Graft-Versus-Host Disease and the Potential Interaction With Fluconazole or Voriconazole
Brief Title: Evaluation of Budesonide and How It Interacts With Antifungal Drugs in People With Gastrointestinal Graft-Versus-Host Disease
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow/Insufficient accrual
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 130197; 13-H-0197
Record Dates: First submitted 2013-09-21; First posted 2013-09-25 (Estimated); Last update posted 2021-03-12 (Actual); Status verified 2020-03

CONDITIONS: Stem Cell Transplantation; Graft vs Host Disease
Keywords: Fluconazole; Graft Versus Host Disease; Voriconazole; Azoles
MeSH Terms: conditions — Graft vs Host Disease | interventions — Budesonide; Fluconazole; Voriconazole; Micafungin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): subjects may be on fluconazole or micafungin at study entry or be on no antifungal prophylaxis.
  Interventions: Drug: Budesonide; Drug: Micafungin
- Cohort 2 (Experimental): subjects are on voriconazole at study entry. Voriconazole will continue throughout days O to 7.
  Interventions: Drug: Voriconazole; Drug: Micafungin
- Cohort 3 (Experimental): subjects are on fluconazole at study entry. Fluconazole will continue throughout days O to 7.
  Interventions: Drug: Fluconazole; Drug: Micafungin

INTERVENTIONS:
Drug: Budesonide — Entocort EC 3 mg given orally three times daily for at least 14 days
  Arms: Cohort 1
Drug: Fluconazole — 400 mg orally once daily for CrCl greater than or equal to 50 ml/min
  Arms: Cohort 3
Drug: Voriconazole — Subjects in Cohort 1 who are not established on voriconazole will receive a loading dose of 400 mg orally every 12 hours for 2 doses, then 200 mg orally every 12 hours
  Arms: Cohort 2
Drug: Micafungin — Micafungin will be dosed as 100 mg as an intravenous infusion once daily at 09:00 for inpatients, and 200 mg to 300 mg as an intravenous infusion administered two to three times weekly for outpatients

SUMMARY:
Background:

The gastrointestinal (GI) tract is commonly affected by acute graft-versus-host disease (aGVHD) and chronic GVHD (cGVHD) in patients who have undergone blood or marrow stem cell transplantation (BMT). Initially, patients are treated with systemic corticosteroids, which produce complete response rates in 35 percent. Although short courses of steroids are preferred to minimize adverse effects, many patients require systemic treatment chronically since GI GVHD can negatively impact quality of life and nutrition status. One option to minimize systemic steroid exposure is by nonabsorbable corticosteroids that act locally on the GI tract.

Budesonide (Entocort EC, AstraZeneca, Wilmington, DE) is an FDA-approved oral topical corticosteroid for the treatment of mild to moderate active Crohn s disease involving the ileum and/or the ascending colon, and for maintenance of clinical remission of mild to moderate Crohn s disease involving the ileum and/or the ascending colon for up to 3 months. It has a high ratio of topical-to-systemic activity with minimally active metabolites, and undergoes extensive first-pass metabolism. Since both intestinal GVHD and Crohn s disease seem to share a similar pathogenic background, budesonide has been used in the BMT setting for GI GVHD, usually in combination with systemic corticosteroids (e.g. methylprednisolone) to improve clinical response and allow for more rapid tapering of systemic corticosteroid doses.

First-pass metabolism is mediated mostly by the cytochrome P450 (CYP450) enzyme system. The liver is the major site of CYP450-mediated metabolism but the enterocytes of the intestinal epithelium are also an important site for drug metabolism. Budesonide undergoes significant metabolism by CYP enzymes with substantial first-pass metabolism. The potential for greater systemic availability of orally administered budesonide exists when it is given concurrently with triazole antifungals, which are commonly prescribed for prophylaxis or treatment of fungal infections after transplantation. Fluconazole and voriconazole are moderate and strong inhibitors of CYP3A4, respectively, and budesonide is a CYP3A4 substrate. Inhibition of CYP3A4 may impair the metabolism of budesonide, resulting in systemic concentrations of budesonide and subsequently, adverse effects such as hyperglycemia. If the presence of fluconazole or voriconazole does impair budesonide s metabolism, then dose adjustments to budesonide may be warranted.

There are no prospective studies evaluating the effects of fluconazole or voriconazole on budesonide s pharmacokinetics in patients who have undergone BMT.

The primary objective of the proposed study is to determine the effects of fluconazole and voriconazole on the trough (Cmin) and peak (Cmax) of budesonide in patients who have undergone BMT and who have GI GVHD.

The primary endpoints are the Cmin and Cmax of budesonide. Secondary endpoints include the Cmin of voriconazole.

Objectives:

The proposed study seeks to determine the effects of fluconazole and voriconazole on the Cminand Cmax of budesonide.

Eligibility:

Adult and pediatric subjects (greater than or equal to 13 years of age and greater than or equal to 49 kg) who are registered to an NCI or NHLBI protocol who have undergone a bone marrow, cord, haplo-cord or peripheral blood stem cell transplantation who have GI GVHD as determined by the medical team and who require treatment with budesonide and are candidates for antifungal therapy are eligible for this study.

Design:

Each subject will serve as his or her own control to minimize the variation in absorption, distribution, metabolism and elimination of oral budesonide that can occur from subject to subject, due to genetic, anatomic or other unidentified differences. For example, genetic polymorphisms of CYP2C19, which is significantly involved in voriconazole s metabolism, could otherwise affect the results of the study (i.e. CYP2C19 poor metabolizers may experience higher voriconazole serum concentrations, which could results in greater CYP3A4 inhibition and higher budesonide exposure). In addition, the longitudinal cohort design of this study will be able to answer the research questions posed with fewer research subjects. Research subjects will be accrued into one of three cohorts depending on the antifungal prophylaxis (or lack thereof) the subject is receiving at study entry and the preference of the medical team for continued antifungal coverage after the initiation of budesonide and systemic corticosteroids. Subjects who are not currently receiving antifungal prophylaxis or who are on fluconazole at baseline are eligible for enrollment in Cohort 1. Subjects in Cohorts 2 and 3 are receiving voriconazole and fluconazole at study entry, respectively. In Cohort 1, if applicable, subjects will stop fluconazole on day -1...

DETAILED DESCRIPTION:
Background:

The gastrointestinal (GI) tract is commonly affected by acute graft-versus-host disease (aGVHD) and chronic GVHD (cGVHD) in patients who have undergone blood or marrow stem cell transplantation (BMT). Initially, patients are treated with systemic corticosteroids, which produce complete response rates in 35 percent. Although short courses of steroids are preferred to minimize adverse effects, many patients require systemic treatment chronically since GI GVHD can negatively impact quality of life and nutrition status. One option to minimize systemic steroid exposure is by nonabsorbable corticosteroids that act locally on the GI tract.

Budesonide (Entocort EC, AstraZeneca, Wilmington, DE) is an FDA-approved oral topical corticosteroid for the treatment of mild to moderate active Crohn s disease involving the ileum and/or the ascending colon, and for maintenance of clinical remission of mild to moderate Crohn s disease involving the ileum and/or the ascending colon for up to 3 months. It has a high ratio of topical-to-systemic activity with minimally active metabolites, and undergoes extensive first-pass metabolism. Since both intestinal GVHD and Crohn s disease seem to share a similar pathogenic background, budesonide has been used in the BMT setting for GI GVHD, usually in combination with systemic corticosteroids (e.g. methylprednisolone) to improve clinical response and allow for more rapid tapering of systemic corticosteroid doses.

First-pass metabolism is mediated mostly by the cytochrome P450 (CYP450) enzyme system. The liver is the major site of CYP450-mediated metabolism but the enterocytes of the intestinal epithelium are also an important site for drug metabolism. Budesonide undergoes significant metabolism by CYP enzymes with substantial first-pass metabolism. The potential for greater systemic availability of orally administered budesonide exists when it is given concurrently with triazole antifungals, which are commonly prescribed for prophylaxis or treatment of fungal infections after transplantation. Fluconazole and voriconazole are moderate and strong inhibitors of CYP3A4, respectively, and budesonide is a CYP3A4 substrate. Inhibition of CYP3A4 may impair the metabolism of budesonide, resulting in systemic concentrations of budesonide and subsequently, adverse effects such as hyperglycemia. If the presence of fluconazole or voriconazole does impair budesonide s metabolism, then dose adjustments to budesonide may be warranted.

There are no prospective studies evaluating the effects of fluconazole or voriconazole on budesonide s pharmacokinetics in patients who have undergone BMT.

The primary objective of the proposed study is to determine the effects of fluconazole and voriconazole on the trough (Cmin) and peak (Cmax) of budesonide in patients who have undergone BMT and who have GI GVHD.

The primary endpoints are the Cmin and Cmax of budesonide. Secondary endpoints include the Cmin of voriconazole.

Objectives:

The proposed study seeks to determine the effects of fluconazole and voriconazole on the Cminand Cmax of budesonide.

Eligibility:

Adult and pediatric subjects (greater than or equal to 13 years of age and greater than or equal to 49 kg) who are registered to an NCI or NHLBI protocol who have undergone a bone marrow, cord, haplo-cord or peripheral blood stem cell transplantation who have GI GVHD as determined by the medical team and who require treatment with budesonide and are candidates for antifungal therapy are eligible for this study.

Design:

Each subject will serve as his or her own control to minimize the variation in absorption, distribution, metabolism and elimination of oral budesonide that can occur from subject to subject, due to genetic, anatomic or other unidentified differences. For example, genetic polymorphisms of CYP2C19, which is significantly involved in voriconazole s metabolism, could otherwise affect the results of the study (i.e. CYP2C19 poor metabolizers may experience higher voriconazole serum concentrations, which could results in greater CYP3A4 inhibition and higher budesonide exposure). In addition, the longitudinal cohort design of this study will be able to answer the research questions posed with fewer research subjects. Research subjects will be accrued into one of three cohorts depending on the antifungal prophylaxis (or lack thereof) the subject is receiving at study entry and the preference of the medical team for continued antifungal coverage after the initiation of budesonide and systemic corticosteroids. Subjects who are not currently receiving antifungal prophylaxis or who are on fluconazole at baseline are eligible for enrollment in Cohort 1. Subjects in Cohorts 2 and 3 are receiving voriconazole and fluconazole at study entry, respectively. In Cohort 1, if applicable, subjects will stop fluconazole on day -1, and may start micafungin on day 0, which will continue through the period off azole prophylaxis if the subject is on systemic corticosteroids (and antifungal prophylaxis is deemed necessary). Voriconazole will be initiated in the evening on day 7. In Cohorts 2 and 3, fluconazole and voriconazole will be discontinued on day 7, and micafungin will be added during the period off azole prophylaxis if the subject is on systemic corticosteroids (and antifungal prophylaxis is deemed necessary). In all three cohorts, a budesonide Cmin and Cmax will be measured both in the presence and absence of concurrent fluconazole or voriconazole therapy. At least a seven day interval will be used between interventions to allow for steady state to occur prior to measurement of budesonide serum concentrations. There is no literature on the interaction between oral budesonide and micafungin, but pharmacokinetic data suggest that micafungin has a low potential to cause drug-drug interactions through inhibition of CYP3A4, and thus it is assumed that micafungin will not significantly affect the Cmin or Cmax of budesonide in this study.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Adult and pediatric subjects (greater than or equal to 13 years of age and greater than or equal to 49 kg)
* Be registered to an NIH protocol that includes bone marrow, cord, haplo-cord or peripheral blood stem cell transplantation
* Have GI GVHD as determined by the medical team that requires treatment with budesonide and systemic corticosteroids (e.g. methylprednisolone or prednisone)
* Be candidates for antifungal therapy
* Liver function tests:

  * Alanine aminotransferase (ALT) must be <5 times the upper limit of normal (ULN)
  * Aspartate aminotransferase (AST) must be <5 times ULN

EXCLUSION CRITERIA:

* Pregnant or breast-feeding
* Prohibited drugs

  --Note: Treatment with corticosteroids and/or immunosuppressants is permitted
* Consumption of grapefruit juice or grapefruit in the past seven days prior to study enrollment
* Inability to take oral medications
* Allergy(ies) to budesonide, fluconazole, micafungin, voriconazole
* ECOG performance status greater than or equal to 4 (adults and children 16 years and older) or Lansky perfomance status less than or equal to 30 (children< 16 years old)
* Psychiatric disorder or mental deficiency that could interfere with the subject s ability to comply with study procedures and requirements
* Inability to provide informed consent
* Major anticipated illness or organ failure whereby the subject s anticipated survival within 2 weeks is unlikely (PI discretion)
* Current documented or suspected invasive fungal infection
* Intensive care unit (ICU) patient
* Child-Pugh Class C hepatic impairment
* AST greater than or equal to 5 times ULN, ALT greater than or equal to 5 times ULN
* Contraindication to an azole as determined by research team
* Body weight < 49 kg at the time of study enrollment

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-02-20 (Actual); Primary Completion 2018-05-10 (Actual); Study Completion 2020-02-26 (Actual)

PRIMARY OUTCOMES:
Cmin and Cmax of budesonide | 2 weeks
  To detect a 2-fold difference in the budesonide Cmax before and after azole administration between study day 7 and day 14 for each cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Hughes, Pharm.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Ross WA, Couriel D. Colonic graft-versus-host disease. Curr Opin Gastroenterol. 2005 Jan;21(1):64-9. PMID 15687887
- [Background] Andree H, Hilgendorf I, Leithaeuser M, Junghanss C, Holzhueter S, Loddenkemper C, Steiner B, Freund M, Wolff D. Enteral budesonide in treatment for mild and moderate gastrointestinal chronic GVHD. Bone Marrow Transplant. 2008 Oct;42(8):541-6. doi: 10.1038/bmt.2008.209. Epub 2008 Jul 21. PMID 18641680
- [Background] Ibrahim RB, Abidi MH, Cronin SM, Lum LG, Al-Kadhimi Z, Ratanatharathorn V, Uberti JP. Nonabsorbable corticosteroids use in the treatment of gastrointestinal graft-versus-host disease. Biol Blood Marrow Transplant. 2009 Apr;15(4):395-405. doi: 10.1016/j.bbmt.2008.12.487. Epub 2009 Feb 10. PMID 19285626
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2013-H-0197.html